CLINICAL TRIAL: NCT04151771
Title: Low-load Blood Flow Restriction Training in COPD
Acronym: LL-BFRT COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-01641; SNCTP000003509 (Other: kofam); 2019-01641 (Other: KEK-ZH)
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: COPD; Muscle Weakness
Keywords: blood flow restriction training; pulmonary rehabilitation; COPD; muscle weakness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LL-BFRT group (Experimental): Participants randomised into intervention group are attending pulmonary rehabilitation in which strengthening exercises of the lower limb are performed using LL-BFRT.
  Interventions: Other: Low-load blood flow restriction training
- Usual pulmonary rehabilitation group (Active Comparator): Participants randomised into control group are attending usual pulmonary rehabilitation as established.
  Interventions: Other: Usual outpatient pulmonary rehabilitation

INTERVENTIONS:
Other: Low-load blood flow restriction training — The intervention group will perform the exercises of the lower limbs using LL-BFRT with an occlusion pressure of 70% of arterial occlusion pressure with low training loads (30% of the 1 repetition maximum).
  Other Names: LL-BFRT
  Arms: LL-BFRT group
Other: Usual outpatient pulmonary rehabilitation — The control group will perform outpatient pulmonary rehabilitation as established.
  Arms: Usual pulmonary rehabilitation group

SUMMARY:
Peripheral muscle weakness is a predominant problem in patients with COPD and treated using exercise training in pulmonary rehabilitation. Despite pulmonary rehabilitation being an effective intervention, muscle strength impairment is a persisting problem in COPD patients. Patients have problems to tolerate the high training loads, which are necessary to develop strength. Low-load blood flow restriction training (LL-BFRT) might therefore be an option to enhance muscular response of patients with COPD to strength training. Up to now, no studies investigating LL-BFRT in respiratory diseases are available.

The primary outcome of this randomized pilot study is knee extensor muscle strength. Secondary, the study will evaluate if LL-BFRT is well tolerated and feasible in COPD patients attending outpatient pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD according to GOLD-guidelines
* Assigned to outpatient pulmonary rehabilitation by the treating physician

Exclusion Criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Non-German speaking (precluding informed consent)
* Acute or recent (within the last 6 weeks) exacerbation of COPD
* Attending a pulmonary rehabilitation program within the last 3 months
* Pregnant patients
* History of thromboembolic event in the lower extremity
* Diagnosis of polyneuropathy
* Resting systolic blood pressure <100 mmHg

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Knee extensor strength | during 12 weeks (24 exercise sessions)
  Between-group difference in total change in isometric muscle strength of the knee extensor muscles, measured by handheld dynamometry in newtonmeter

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kohlbrenner D, Kuhn M, Manettas A, Aregger C, Peterer M, Greco N, Sievi NA, Clarenbach C. Low-load blood flow restriction strength training in patients with COPD: a randomised single-blind pilot study. Thorax. 2024 Mar 15;79(4):340-348. doi: 10.1136/thorax-2023-220546. PMID 38129116